CLINICAL TRIAL: NCT06645106
Title: Offering Routine and Rapid Point of Care (POC) Syphilis Testing in Pregnant Patients Presenting to the Emergency Department
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Irene Stafford, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MS-24-0505
Record Dates: First submitted 2024-10-07; First posted 2024-10-16 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Syphilis
Keywords: syphilis diagnostic testing; pregnancy
MeSH Terms: conditions — Syphilis | interventions — Surgical Instruments; Syphilis Serodiagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Rapid Point of Care (POC) Syphilis testing (Experimental)
  Interventions: Device: Rapid Point of Care (POC) Syphilis testing

INTERVENTIONS:
Device: Rapid Point of Care (POC) Syphilis testing — Participants will undergo the point of care (POC) FDA cleared syphilis health check (SHC) POC test by a research staff using 50 microliters or 1-3 drops of whole blood via finger stick. The analyzer is handheld, and all testing equipment is temperature stable and does not need refrigeration. The SHC-Syphilis results will be available within 10 minutes of receipt given the published turnaround time to results of 15 minutes per package insert and will be recorded as a research note in the electronic medical record (EMR) while the provider assigned to the patient and the Houston Health Department will be notified of results and further treatment will be done if results are positive.

SUMMARY:
The purpose of this study is to offer routine lab-based and rapid point of care (POC) syphilis diagnostic testing in the emergency department (ED) and obstetrical (OB) triage , thereby increasing screening and treatment initiation for pregnant patients without prenatal care or with no documented syphilis results during the index pregnancy in other to increase rates of full treatment to determine if the implementation of a robust linkage to care program for pregnant patients with positive rapid POC results will more likely result in complete treatment for all stages of syphilis and adherence to recommended maternal and newborn longitudinal follow up and to assess factors that contribute to treatment completion after implementation of the intervention will also be analyzed to tailor efforts targeting social and healthcare navigation factors that affect health equity; including poverty, insurance, health literacy and others.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individuals that are seeking care at University of Texas, Memorial Herman and Lyndon B Johnson sites ED or obstetrical triage units.
* No Prenatal care during index pregnancy
* No documented syphilis result during the index pregnancy

Exclusion Criteria:

* Pregnant individuals with documented care and syphilis results in the index pregnancy for specific trimester as mandated by Texas law

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-01-06 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients without prenatal care during the index pregnancy who received full treatment for all stages of syphilis | within 1 week of presentation until the time of delivery
Percentage of patients with no documented syphilis test during the index pregnancy who received full treatment for all stages of syphilis | within 1 week of presentation until the time of delivery

SECONDARY OUTCOMES:
The percentage of patients who adhere to recommended maternal and newborn longitudinal follow up | within 1 week of presentation until the time of delivery
The percentage of patients who adhere to recommended maternal and newborn longitudinal follow up | at time of postpartum (upto 15 months after delivery)
Percentage of participants that are married on completion of syphilis treatment | from presentation to delivery
Percentage of participants that have health insurance on completion of syphilis treatment | from presentation to delivery
Percentage of participants that have psychiatric problems on completion of syphilis treatment | from presentation to delivery
Percentage of participants that show substance abuse including alcohol on completion of syphilis treatment | from presentation to delivery
Percentage of participants that have unstable housing on completion of syphilis treatment | from presentation to delivery
Percentage of participants that have transportation on completion of syphilis treatment | from presentation to delivery
Percentage of participants that experience intimate partner violence on completion of syphilis treatment | from presentation to delivery
number of prenatal care visits on completion of syphilis treatment | from presentation to delivery
Percentage of participants that are married on completion of syphilis treatment | at time of postpartum (upto 15 months after delivery)
Percentage of participants that have health insurance on completion of syphilis treatment | at time of postpartum (upto 15 months after delivery)
Percentage of participants that have psychiatric problems on completion of syphilis treatment | at time of postpartum (upto 15 months after delivery)
Percentage of participants that show substance abuse including alcohol on completion of syphilis treatment | at time of postpartum (upto 15 months after delivery)
Percentage of participants that have unstable housing on completion of syphilis treatment | at time of postpartum (upto 15 months after delivery)
Percentage of participants that have transportation on completion of syphilis treatment | at time of postpartum (upto 15 months after delivery)
Percentage of participants that experience intimate partner violence on completion of syphilis treatment | at time of postpartum (upto 15 months after delivery)
number of prenatal care visits on completion of syphilis treatment | at time of postpartum (upto 15 months after delivery)
Number of birth parents that have reinfection | from presentation to delivery
Number of birth parents that have reinfection | at time of postpartum (upto 15 months after delivery)
Number of neonates that have congenital syphilis | from presentation to delivery
Number of neonates that have congenital syphilis | at time of postpartum (upto 15 months after delivery)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Stafford, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No